CLINICAL TRIAL: NCT02034019
Title: Phase 3 Study Evaluating Safety and Efficacy of OTX-DP for Treatment of Ocular Inflammation and Pain After Cataract Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Ocular Therapeutix, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: OTX-13-002
Record Dates: First submitted 2014-01-09; First posted 2014-01-13 (Estimated); Results first posted 2020-01-31 (Actual); Last update posted 2020-01-31 (Actual); Status verified 2020-01

CONDITIONS: Post Ocular Surgical Inflammation and Pain
MeSH Terms: conditions — Pain | interventions — Dexamethasone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- OTX-DP (Dexamethasone Punctum Plug) (Active Comparator): Resorbable hydrogel drug delivery vehicle containing dexamethasone
  Interventions: Drug: Dexamethasone; Drug: Punctum Plug
- PVPP (Placebo Punctum Plug) (Placebo Comparator): Resorbable hydrogel drug delivery vehicle containing no drug
  Interventions: Drug: Punctum Plug

INTERVENTIONS:
Drug: Dexamethasone
  Arms: OTX-DP (Dexamethasone Punctum Plug)
Drug: Punctum Plug

SUMMARY:
To evaluate the safety and efficacy of OTX-DP as a sustained release drug (dexamethasone) depot when placed in the canaliculus of the eyelid for the treatment of post-surgical inflammation and pain in subjects who have undergone cataract extraction with intra-ocular lens implantation.

ELIGIBILITY:
Inclusion Criteria:

* Has a cataract and is expected to undergo clear corneal cataract surgery with phacoemulsification and implantation of a posterior chamber intraocular lens
* Has a potential post-operative pinhole corrected Snellen VA of at least 20/200 or better in both eyes

Exclusion Criteria:

* Any intraocular inflammation in the study eye present during the screening slit lamp examination
* Score greater than "0" on the Ocular Pain Assessment in the study eye at Screening
* Any intraocular inflammation in the study eye present during the screening slit lamp examination

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 247 (Actual)
Dates: Start 2014-02; Primary Completion 2014-12 (Actual); Study Completion 2015-02 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Project Manager, Study Director — Ocular Therapeutix
Locations (1):
- Texan Eye / Keystone Research, Ltd., Austin, Texas, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: One subject inadvertently received PVPP instead of OTX-DP, as they had been randomized. This subject was followed safety but not included in the PP analysis.
Groups:
- OTX-DP (Dexamethasone Punctum Plug): Resorbable hydrogel drug delivery vehicle containing dexamethasone
  Dexamethasone
  Punctum Plug
- PVPP (Placebo Punctum Plug): Resorbable hydrogel drug delivery vehicle containing no drug
  Punctum Plug
Period: Overall Study
Arm/Group | OTX-DP (Dexamethasone Punctum Plug) | PVPP (Placebo Punctum Plug)
Started | 164 | 83
Completed | 163 | 81
Not Completed | 1 | 2

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | OTX-DP (Dexamethasone Punctum Plug) | PVPP (Placebo Punctum Plug) | Total
Number analyzed (Participants) | 164 | 83 | 247
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 56 | 16 | 72
  >=65 years | 108 | 67 | 175
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 103 | 44 | 147
  Male | 61 | 39 | 100

OUTCOME MEASURES:

1. Primary Outcome: Absence of Cells in Anterior Chamber of the Study Eye
Time Frame: Day 14
Measure: Count of Participants; unit: Participants
Arm/Group | OTX-DP (Dexamethasone Punctum Plug) | PVPP (Placebo Punctum Plug)
Number analyzed (Participants) | 164 | 83
Participants | 54 | 12

2. Primary Outcome: Absence of Pain in Study Eye
Time Frame: Day 8
Measure: Count of Participants; unit: Participants
Arm/Group | OTX-DP (Dexamethasone Punctum Plug) | PVPP (Placebo Punctum Plug)
Number analyzed (Participants) | 164 | 83
Participants | 131 | 36

ADVERSE EVENTS:
Description: One subject was inadvertently treated with PVPP instead of OTX-TP, as they had been randomized. This subject was not included in the PP, but was followed for safety.
Arm/Group | OTX-DP (Dexamethasone Punctum Plug) | PVPP (Placebo Punctum Plug)
Serious Adverse Events (participants affected / at risk) | 0/162 | 1/84
Other Adverse Events (participants affected / at risk) | 37/162 | 31/84
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-DP (Dexamethasone Punctum Plug) (N=162) | PVPP (Placebo Punctum Plug) (N=84)
hypopyon (Eye disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | OTX-DP (Dexamethasone Punctum Plug) (N=162) | PVPP (Placebo Punctum Plug) (N=84)
inflammation (Eye disorders) | 37 (47) | 31 (38)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other